CLINICAL TRIAL: NCT06067191
Title: A RANDOMISED, PHASE 1B, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY TO EVALUATE THE SAFETY, PHARMACOKINETICS, AND ANTIVIRAL ACTIVITY OF RV299 AGAINST RESPIRATORY SYNCYTIAL VIRUS IN THE VIRAL CHALLENGE MODEL
Brief Title: Safety, Pharmacokinetics,and Antiviral Activity of RV299 Against Respiratory Syncytical Virus (RSV)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: REVD002; C5251002 (Other: Alias Study Number)
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-07

CONDITIONS: Respiratory Syncytial Virus (RSV)
Keywords: Anti-viral; Challenge

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): spray-dried dispersion (SDD) for Oral Suspension
  Interventions: Drug: RV299
- Placebo (Placebo Comparator): spray-dried dispersion (SDD) for Oral Suspension
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RV299 — Oral Suspension
  Arms: Active
Drug: Placebo — matching placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to learn about the safety, pharmacokinetics and antiviral activity of the study medicine (RV299) for the potential treatment of respiratory syncytial virus (RSV). RSV is a highly contagious virus that can lead to serious lung infections in patients with reduced ability to fight infection. Most vulnerable populations include babies, the elderly and patients that have received a bone marrow transplant.

DETAILED DESCRIPTION:
This study is seeking healthy participants who are:

Healthy adult male and female participants aged between 18 to 55 years, with a total body weight ≥50 kg and body mass index (BMI) ≥18 kg/m2 and ≤35kg/m2 and who have been screened to be sero-suitable for infection with the RSV-A Memphis 37b virus challenge virus.

A total of 80 participants is planned: 40 participants on RV299 and 40 participants on placebo.

The study is divided into 3 phases:

* Screening phase: from Day -90 to Day-3 pre-human viral challenge (HVC).
* Inpatient phase: Participants will be resident in the quarantine unit for approximately 15 days (from Day -2 to Day 12).

  * Post RSV-A Memphis 37b virus inoculation on Day 0, participants will be randomized to receive RV299 or matched placebo.
  * Administration of RV299 or placebo will be twice daily (~12 hours interval) for 5 consecutive days and will start on confirmation of RSV infection.
* Outpatient phase: Day 28 (±3 days)

ELIGIBILITY:
Inclusion Criteria:

* Total body weight >= 50 kg and body mass index (BMI) >=18 kg/m2 and <=35 kg/m2
* in good health with no history, or current evidence of clinically significant medical condition of laboratory, ECG or vital sign abnormality
* Sero suitable for challenge virus

Exclusion Criteria:

* History of or currently active symptoms or signs suggestive of upper or lower respiratory tract infection within 4 weeks prior to first study visit
* Any history or evidence of any clinically significant or currently active cardiovascular, respiratory, dermatological, gastrointestinal, endocrinological, haematological, hepatic, immunological (including immunosuppression),metabolic, urological, renal, neurological, or psychiatric disease and/or other major disease
* females who are breastfeeding or have been pregnant within 6 months prior to the study or have a positive pregnancy test
* Lifetime history of anaphylaxis and/or a lifetime history of severe allergic reaction
* Any significant abnormality altering the anatomy of the nose in a substantial way
* Any clinically significant history of epistaxis (large nosebleeds)
* Any nasal or sinus surgery within 3 months of first study visit
* Evidence of vaccinations within 4 weeks of Day 0
* Receipt of blood or blood products, or loss of 550 mL or more blood within last 3 months
* Receipt of 3 or more investigational drug within last 12 months
* Prior inoculation with a virus from the same virus-family as the challenge
* Prior participation in another HVC study with a respiratory virus in last 3 months
* Use or anticipated use during the conduct of the study of protocol specified concomitant medications
* Systemic antiviral administration within 4 weeks of viral challenge
* Confirmed positive test for drugs of abuse
* History or presence of alcohol addiction, or excessive use of alcohol
* A forced expiratory volume in 1 second (FEV1) <80%
* Positive HIV, hepatitis B virus, or hepatitis C virus test
* Presence of fever upto 2 days prior to Day 0.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=REVD002

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 82 healthy participants were enrolled in the study and received Respiratory Syncytial Virus (RSV) - A Memphis 37b virus inoculation (challenge agent) intranasally on Day 0. Three participants withdrew from study (2 withdrew consent and 1 not randomized because of influenza infection) before randomization and a total of 79 participants were randomized in the study.
Groups:
- RV299: Participants were administered an oral suspension of 65 milligrams (mg) RV299 twice daily at an interval of approximately 12 hours for 5 consecutive days from Day 2 following confirmation of RSV infection. Participants without a positive result for RSV infection were administered RV299 from Day 5.
- Placebo: Participants were administered an oral suspension of placebo twice daily at an interval of approximately 12 hours for 5 consecutive days from Day 2 following confirmation of RSV infection. Participants without a positive result for RSV infection were administered placebo from Day 5.
Period: Overall Study
Arm/Group | RV299 | Placebo
Started | 39 | 40
Completed | 39 | 39
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population consisted of all randomized participants who received challenge virus and at least one dose of investigational medicinal product (IMP).
Groups:
- Total: Total of all reporting groups
Arm/Group | RV299 | Placebo | Total
Number analyzed (Participants) | 39 | 40 | 79
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.7 (6.21) | 26.2 (7.29) | 25.9 (6.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 22 | 23 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 30 | 30 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) for RSV-A Memphis 37b Viral Load Determined by Quantitative Real Time Reverse Transcription Polymerase Chain Reaction (qRT-PCR)
Description: Area under the curve (AUC) for RSV viral load measured in nasal washes by qRT-PCR in participants inoculated with RSV-A Memphis 37b, from initial administration of IMP up to the morning of Day 12 (Quarantine discharge) was presented in this outcome measure.
Time Frame: From initial administration of IMP up to the morning of quarantine discharge (up to Day 12)
Population: Intent-to-Treat Infected (ITT-I) Population consisted of all randomized participants who received challenge virus and at least 1 dose of IMP and met the criterion for RSV infection.
Measure: Mean (Standard Deviation); unit: Hours*log10 copies per milliliter
Arm/Group | RV299 | Placebo
Number analyzed (Participants) | 23 | 29
Hours*log10 copies per milliliter | 350.99 (289.79) | 616.97 (374.143)
Statistical Analysis 1: Comparison: RV299 vs Placebo; Test type: Other; p = 0.0009, ANCOVA; Difference in Least Square Mean = -312.28, 95% CI 2-sided [-489.17 to -135.38] — Analysis was performed using ANCOVA with treatment group as a fixed effect and baseline viral load as the covariate

2. Secondary Outcome: Peak Viral Load of RSV Determined by qRT-PCR
Description: Peak viral load of RSV as defined by the maximum viral load determined by qRT-PCR measurements in nasal samples starting from initial administration of IMP up to planned discharge from quarantine was reported in this outcome measure.
Time Frame: From initial administration of IMP up to planned discharge from quarantine (Up to Day 12)
Population: ITT-I Population consisted of all randomized participants who received challenge virus and at least 1 dose of IMP and met the criterion for RSV infection.
Measure: Mean (Standard Deviation); unit: Log10 copies per milliliter
Arm/Group | RV299 | Placebo
Number analyzed (Participants) | 23 | 29
Log10 copies per milliliter | 5.01 (1.968) | 6.23 (1.735)
Statistical Analysis 1: Comparison: RV299 vs Placebo; Test type: Other; p = 0.0047, ANCOVA; Difference in Least Square Mean = -1.45, 95% CI 2-sided [-2.43 to -0.47] — Analysis was performed using ANCOVA with treatment group as a fixed effect and baseline viral load as the covariate

3. Secondary Outcome: Time to Confirmed Negative Test by qRT-PCR Measurement Starting From Initial Administration of Investigational Medicinal Product (IMP) to First Confirmed Undetectable Assessment After Peak Measure
Description: The time from the first administration of IMP to the first confirmed negative qRT-PCR test after the peak qRT-PCR measurement was calculated as: Date and time of first confirmed negative test after peak qRT-PCR measurement minus Date and time of first IMP administration. A negative test was defined as two consecutive 'Not Detected' results in the qRT-PCR test. The peak qRT-PCR was defined as the highest viral load value obtained by a participant after their first administration of IMP. Participants without a confirmed undetectable assessment after their peak, were censored at their last detected qRT-PCR assessment.
Time Frame: From first administration of IMP to the first confirmed negative qRT-PCR test or censoring date (up to Day 12)
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | RV299 | Placebo
Number analyzed (Participants) | 23 | 29
Days | 4.2 [2.0 to 6.5] | 8.5 [6.0 to 9.0]
Statistical Analysis 1: Comparison: RV299 vs Placebo; Test type: Other; p < 0.0001, Log Rank

4. Secondary Outcome: Time to Confirmed Negative Test by qRT-PCR Measurement Starting From Peak qRT-PCR After Initial Administration of IMP to First Confirmed Undetectable Assessment After Peak Measure
Description: The time from the peak qRT-PCR measurement after administration of IMP to the first confirmed negative qRT-PCR test was calculated as (Date and time of first confirmed negative test after peak qRT-PCR measurement minus Date and time of peak qRT-PCR measurement). A negative test was defined as two consecutive 'Not Detected' results in the qRT-PCR test. The peak qRT-PCR was defined as the highest viral load value obtained by a participant after their first administration of IMP. Participants without a confirmed undetectable assessment after their peak, were censored at their last detected qRT-PCR assessment.
Time Frame: From peak qRT-PCR measurement to the first confirmed negative qRT-PCR test or censoring date (up to Day 12)
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | RV299 | Placebo
Number analyzed (Participants) | 23 | 29
Days | 2.5 [1.5 to 4.5] | 5.0 [2.5 to NA] — Upper limit of interquartile range could not be calculated due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: RV299 vs Placebo; Test type: Other; p = 0.0051, Log Rank

5. Secondary Outcome: Time to Peak qRT-PCR Starting From Initial Administration of IMP
Description: The time to the peak qRT-PCR measurement starting from the initial administration of IMP was calculated as: Date and time of peak qRT-PCR measurement minus Date and time of first IMP administration. The peak qRT-PCR was defined as the highest viral load value obtained by a participant after their first administration of IMP.
Time Frame: From first administration of IMP to peak qRT-PCR measurement (up to Day 12)
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | RV299 | Placebo
Number analyzed (Participants) | 23 | 29
Days | 1.5 [0.5 to 2.0] | 1.5 [1.5 to 4.0]
Statistical Analysis 1: Comparison: RV299 vs Placebo; Test type: Other; p = 0.0077, Log Rank

6. Secondary Outcome: Area Under the Viral Load-Time Curve (VL-AUC) for RSV-A Memphis 37b Determined by Viral Culture
Description: Area under the viral load-time curve (VL-AUC) of RSV challenge virus as determined by viral culture on nasal samples, starting at initial administration of IMP up to planned discharge from quarantine was reported in this outcome measure.
Time Frame: From initial administration of IMP up to planned discharge from quarantine (up to Day 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours*log10 plaque forming units/mL
Arm/Group | RV299 | Placebo
Number analyzed (Participants) | 23 | 29
Hours*log10 plaque forming units/mL | 106.48 (133.187) | 212.51 (170.700)
Statistical Analysis 1: Comparison: RV299 vs Placebo; Test type: Other; p = 0.0268, ANCOVA; Difference in Least Square Mean = -87.40, 95% CI 2-sided [-164.30 to -10.49] — Analysis was performed using ANCOVA with treatment group as a fixed effect and baseline viral load as the covariate

7. Secondary Outcome: Peak Viral Load of RSV Determined by Viral Culture
Description: Peak viral load of RSV as defined by the maximum viral load determined by viral culture measurements in nasal samples starting from initial administration of IMP up to planned discharge from quarantine was reported in this outcome measure.
Time Frame: From initial administration of IMP up to planned discharge from quarantine (up to Day 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 plaque forming units/mL
Arm/Group | RV299 | Placebo
Number analyzed (Participants) | 23 | 29
Log10 plaque forming units/mL | 2.43 (2.030) | 3.63 (2.285)
Statistical Analysis 1: Comparison: RV299 vs Placebo; Test type: Other; p = 0.0865, ANCOVA; Difference in Least Square Mean = -0.99, 95% CI 2-sided [-2.13 to 0.15] — Analysis was performed using ANCOVA with treatment group as a fixed effect and baseline viral load as the covariate

8. Secondary Outcome: Time to Confirmed Negative Test by Viral Culture Measurement Starting From at Initial Administration of IMP to First Confirmed Undetectable Assessment After Peak Measure
Description: Time to confirmed negative test by viral culture measurements in nasal samples from initial administration of IMP up to first confirmed negative viral culture measurement after the peak viral culture measurement was calculated as: Date and time of first confirmed negative test after peak viral culture measurement minus Date and time of first IMP administration. A negative test was defined as two consecutive 'Not Detected' results in the viral culture test. The peak viral culture measurement was defined as the highest viral load value obtained by a participant after their first administration of IMP. Participants who did not have a confirmed undetectable assessment after their peak viral culture measurement after first administration of IMP were censored at their last detectable assessment.
Time Frame: From initial administration of IMP up to first confirmed undetectable assessment or censoring date (up to Day 12)
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | RV299 | Placebo
Number analyzed (Participants) | 23 | 29
Days | 3.2 [2.5 to 3.8] | 5.0 [3.6 to 6.0]
Statistical Analysis 1: Comparison: RV299 vs Placebo; Test type: Other; p = 0.0008, Log Rank

9. Secondary Outcome: Time to Confirmed Negative Test by Viral Culture Measurement Starting From Peak Viral Culture After Initial Administration of IMP to First Confirmed Undetectable Assessment After Peak Measure
Description: The time from the peak viral culture measurement after administration of IMP to the first confirmed negative viral culture measurement was calculated in days as: Date of and time first confirmed negative test minus Date and time of peak qRT-PCR measurement. A negative test was defined as two consecutive 'Not Detected' results in the viral culture test. The peak viral culture measurement was defined as the highest viral load value obtained by a participant after their first administration of IMP. Participants who did not have a confirmed undetectable assessment after their peak viral culture measurement after first administration of IMP were censored at their last detectable assessment.
Time Frame: From peak qRT-PCR measurement to first confirmed undetectable assessment or censoring date (up to Day 12)
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | RV299 | Placebo
Number analyzed (Participants) | 23 | 29
Days | 1.3 [0.7 to 2.5] | 1.6 [1.0 to 2.0]
Statistical Analysis 1: Comparison: RV299 vs Placebo; Test type: Other; p = 0.8579, Log Rank

10. Secondary Outcome: Area Under the Curve Over Time of Total Clinical Symptoms as Measured From 10 Symptoms Within the Graded Symptom Scoring System
Description: Area under the Curve over Time of Total Clinical Symptoms (TSS-AUC) as measured from 10 symptoms within Graded Symptom Scoring System Collected 3 Times Daily Starting at Initial Administration up to Planned Discharge from Quarantine. TSS (from 10 items of the 13-item symptom diary card) was used to calculate the AUC, from the assessment nearest to the time of the first administration of IMP until Day 12. Following types of symptoms were recorded on symptom diary cards: Upper Respiratory Tract (URT): runny nose, stuffy nose, sore throat, sneezing, earache; Lower Respiratory Tract (LRT): cough, shortness of breath; Systemic: headache, malaise, muscle/joint ache/stiffness. Each symptom was recorded on a grading scale of 0 to 3 (or 0 to 4 for the Shortness of Breath symptom), higher scores = greater severity of symptoms. Total symptom score was calculated as sum of the 10 observed symptom grade values and ranged from 0 to 31, where higher scores indicated more severe symptoms.
Time Frame: From initial administration of IMP (before or after administration) up to planned discharge from quarantine (up to Day 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours*score
Arm/Group | RV299 | Placebo
Number analyzed (Participants) | 23 | 29
Hours*score | 180.77 (242.274) | 240.94 (224.439)
Statistical Analysis 1: Comparison: RV299 vs Placebo; Test type: Other; p = 0.0658, ANCOVA; Difference in Least Square Mean = -93.95, 95% CI 2-sided [-194.26 to 6.36] — Analysis was performed using ANCOVA with treatment group as a fixed effect and baseline viral load as the covariate

11. Secondary Outcome: Area Under the Curve Over Time of Total Clinical Symptoms Change From Baseline (TSS-AUC-CFB) as Measured From 10 Symptoms Within the Graded Symptom Scoring System
Description: Area under the curve over time of total clinical symptoms change from baseline (TSS-AUC-CFB) as measured from 10 symptoms within the graded symptom scoring system collected 3 times daily starting at initial administration of IMP up to planned discharge from quarantine (Day 12, am). The following types of symptoms were recorded: Upper Respiratory Tract (URT): runny nose, stuffy nose, sore throat, sneezing, earache; Lower Respiratory Tract (LRT): cough, shortness of breath; Systemic: headache, malaise, muscle/joint ache/stiffness. Each symptom was recorded on a grading scale of 0 to 3 (or 0 to 4 for the Shortness of Breath symptom), where higher scores indicated greater severity of symptoms. TSS was calculated as sum of the 10 observed symptom grade values and ranged from 0 to 31, where higher scores indicated more severe symptoms. The AUC calculation was based on the available non-missing calculated total symptom scores between the start and end of the defined AUC time.
Time Frame: Baseline (assessment nearest to the time of the first administration of IMP) up to Day 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours*score
Arm/Group | RV299 | Placebo
Number analyzed (Participants) | 23 | 29
Hours*score | -17.23 (202.602) | 103.75 (212.465)
Statistical Analysis 1: Comparison: RV299 vs Placebo; Test type: Other; p = 0.0658, ANCOVA; Difference in Least Square Mean = -93.95, 95% CI 2-sided [-194.26 to 6.36] — Analysis was performed using ANCOVA with treatment group as a fixed effect and baseline viral load as the covariate

12. Secondary Outcome: Overall Peak Total Clinical Symptoms (TSS) Score
Description: Peak total clinical symptoms (TSS) as measured from 10 symptoms within the graded symptom scoring system collected 3 times daily starting from initial administration of IMP up to planned discharge from quarantine. The following types of symptoms were recorded: Upper Respiratory Tract (URT): runny nose, stuffy nose, sore throat, sneezing, earache; Lower Respiratory Tract (LRT): cough, shortness of breath; Systemic: headache, malaise, muscle/joint ache/stiffness. Each symptom was recorded on a grading scale of 0 to 3 (or 0 to 4 for the Shortness of Breath symptom), where higher scores indicated greater severity of symptoms. The total symptom score was calculated as sum of the 10 observed symptom grade values and ranged from 0 to 31, where higher scores indicated more severe symptoms. The overall peak score was defined as the highest scoring symptom diary card observed from the first administration of IMP until quarantine discharge.
Time Frame: as for outcome 10
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | RV299 | Placebo
Number analyzed (Participants) | 23 | 29
Units on a scale | 3.30 (2.835) | 3.90 (3.063)
Statistical Analysis 1: Comparison: RV299 vs Placebo; Test type: Other; p = 0.2030, ANCOVA; Difference in Least Square Mean = -0.93, 95% CI 2-sided [-2.38 to 0.52] — Analysis was performed using ANCOVA with treatment group as a fixed effect and baseline viral load as the covariate

13. Secondary Outcome: Individual Maximum Daily Peak Symptom Score
Description: Individual maximum daily sum of symptom score from initial administration of IMP up to planned discharge from quarantine. The following types of symptoms were recorded: Upper Respiratory Tract (URT): runny nose, stuffy nose, sore throat, sneezing, earache; Lower Respiratory Tract (LRT): cough, shortness of breath; Systemic: headache, malaise, muscle/joint ache/stiffness. Each symptom was recorded on a grading scale of 0 to 3 (or 0 to 4 for the Shortness of Breath symptom), where higher scores indicated greater severity of symptoms. The total symptom score was calculated as sum of the 10 observed symptom grade values and ranged from 0 to 31, where higher scores indicated more severe symptoms. The highest total symptom score recorded on each day, across the three assessments was reported in this outcome measure. The peak daily score was defined as the highest scoring symptom diary card observed on each day from the first administration of IMP until quarantine discharge.
Time Frame: Day 0, Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8 and Day 9 (days relative to first administration of IMP)
Population: ITT-I Population consisted of all randomized participants who received challenge virus and at least 1 dose of IMP and met the criterion for RSV infection. Here, 'Number Analyzed' signifies participants evaluable for the specified timepoints.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | RV299 | Placebo
Number analyzed (Participants) | 23 | 29
Units on a scale
  Day 0 | 2.1 (2.32) | 1.2 (1.70)
  Day 1 | 2.0 (2.70) | 1.8 (2.12)
  Day 2 | 1.9 (2.73) | 3.0 (3.01)
  Day 3 | 1.9 (2.83) | 2.6 (2.54)
  Day 4 | 1.1 (1.71) | 2.1 (2.17)
  Day 5 | 0.7 (1.27) | 1.6 (2.11)
  Day 6 | 0.6 (1.12) | 1.0 (1.86)
  Day 7: number analyzed (Participants) | 14 | 16
  Day 7 | 0.6 (1.16) | 1.1 (1.53)
  Day 8: number analyzed (Participants) | 5 | 13
  Day 8 | 1.0 (1.22) | 0.4 (0.51)
  Day 9: number analyzed (Participants) | 2 | 2
  Day 9 | 0.0 (0.0) | 0.0 (0.0)

14. Secondary Outcome: Time to Symptom Resolution Starting at Initial Administration of IMP to 24 Hours Symptom Free
Description: Symptom resolution was defined as a participant scoring 0 for the total symptom score for a 24-hour period (e.g., a minimum of three consecutive symptom diary cards, each with a score of 0) after their peak symptom score. The time from the assessment at the time of the first administration of IMP until symptom resolution was calculated as: Date and time of symptom resolution minus Date and time of assessment at IMP administration. If the peak symptom score occurred on more than one day then the first occurrence was selected. Participants who did not record 24 hours symptom free after their highest total symptom score during the quarantine period were censored at their last assessment.
Time Frame: From first administration of IMP until time of symptom resolution or censoring date (up to Day 12)
Population: ITT-I Population consisted of all randomized participants who received challenge virus and at least 1 dose of IMP and met the criterion for RSV infection. Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | RV299 | Placebo
Number analyzed (Participants) | 19 | 25
Days | 3.99 [1.45 to 6.65] | 6.40 [4.48 to 7.99]

15. Secondary Outcome: Time to Symptom Resolution Starting at Peak Symptoms After Initial Administration to 24 Hours Symptom Free
Description: Symptom resolution was defined as a participant scoring 0 for the total symptom score for a 24-hour period (e.g., a minimum of three consecutive symptom diary cards, each with a score of 0) after their peak symptom score. The time from the highest total symptom score following administration of IMP until symptom resolution was calculated as: Date and time of symptom resolution minus Date and time of highest total symptom score. If the peak symptom score occurred on more than one day then the first occurrence was selected. Participants who did not record 24 hours symptom free after their highest total symptom score during the quarantine period were censored at their last assessment.
Time Frame: From time of highest total symptom score until time of symptom resolution or censoring date (up to Day 12)
Population: as for outcome 14
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | RV299 | Placebo
Number analyzed (Participants) | 19 | 25
Days | 1.44 [0.67 to 3.66] | 3.67 [2.37 to 4.64]

16. Secondary Outcome: Time to Peak Symptom Score From Initial Administration of IMP
Description: Time to peak as measured from 10 symptoms within the graded daily symptom scoring system starting from initial administration of IMP to the time of peak daily symptom score. If the peak symptom score occurred on more than one day then the first occurrence was selected. Participants were censored at their last assessment if they did not record any symptoms during the quarantine period.
Time Frame: From first dose of IMP until time of highest total symptom score or censoring date (Up to Day 12)
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | RV299 | Placebo
Number analyzed (Participants) | 23 | 29
Days | 1.61 [0.42 to 4.63] | 2.74 [1.99 to 3.97]

17. Secondary Outcome: Total Weight of Mucus Produced Starting at Initial Administration of IMP up to Planned Discharge From Quarantine
Description: Total weight of nasal mucus was calculated as the sum of mucus weights taken from the assessment at the time of the first administration of IMP (prior to or after dosing, depending on whether dosed in the morning or evening) to morning of Day 12 (Quarantine discharge).
Time Frame: From first administration of IMP up to planned discharge from quarantine (up to Day 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | RV299 | Placebo
Number analyzed (Participants) | 23 | 29
Grams | 7.49 (14.516) | 16.23 (21.850)

18. Secondary Outcome: Total Number of Tissues Used by Participants Starting At Initial Administration of IMP up to Planned Discharge From Quarantine
Description: Total number of tissues was counted from the assessment at the time of the first dose of IMP (prior to or after dosing, depending on whether dosed in the morning or evening) to morning of Day 12 (Quarantine discharge).
Time Frame: From first administration of IMP up to planned discharge from quarantine (up to Day 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Tissues
Arm/Group | RV299 | Placebo
Number analyzed (Participants) | 23 | 29
Tissues | 14.09 (21.067) | 28.17 (33.078)

19. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An adverse event was defined as any untoward medical occurrence in clinical study participants administered a pharmaceutical product. An AE did not necessarily have a causal relationship with the study intervention. An SAE was defined as any untoward medical occurrence that, at any dose: resulted in death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, was a congenital anomaly/birth defect or important medical event.
Time Frame: From first dose of IMP until end of follow-up visit (up to Day 28)
Population: Safety analysis population was defined as all randomized participants who received challenge virus and at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | RV299 | Placebo
Number analyzed (Participants) | 39 | 40
Participants
  Adverse Event | 12 | 12
  Serious Adverse Event | 0 | 0

20. Secondary Outcome: Number of Participants With AEs Related to Viral Challenge
Description: An Adverse Event was defined as any untoward medical occurrence in clinical study participants administered a pharmaceutical product. An AE did not necessarily have a causal relationship with the study intervention. Number of participants with AEs possibly, probably or definitely related to viral challenge agents were reported by preferred terms in this outcome measure.
Time Frame: From viral challenge on Day 0 up to end of follow-up (Day 28)
Population: Safety analysis population was defined as all randomised participants who received challenge virus and at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | RV299 | Placebo
Number analyzed (Participants) | 39 | 40
Participants
  Headache (Possibly Related) | 2 | 0
  Headache (Probably Related) | 0 | 1
  Headache (Definitely Related) | 0 | 0
  Ageusia (Possibly Related) | 0 | 1
  Ageusia (Probably Related) | 0 | 0
  Ageusia (Definitely Related) | 0 | 0
  Anosmia (Possibly Related) | 0 | 1
  Anosmia (Probably Related) | 0 | 0
  Anosmia (Definitely Related) | 0 | 0
  Syncope (Possibly Related) | 0 | 0
  Syncope (Probably Related) | 0 | 0
  Syncope (Definitely Related) | 0 | 0
  Nausea (Possibly Related) | 0 | 0
  Nausea (Probably Related) | 0 | 0
  Nausea (Definitely Related) | 0 | 0
  Abdominal distension (Possibly Related) | 0 | 0
  Abdominal distension (Probably Related) | 0 | 0
  Abdominal distension (Definitely Related) | 0 | 0
  Diarrhoea (Possibly Related) | 0 | 0
  Diarrhoea (Probably Related) | 0 | 0
  Diarrhoea (Definitely Related) | 0 | 0
  Mouth ulceration (Possibly Related) | 1 | 0
  Mouth ulceration (Probably Related) | 0 | 0
  Mouth ulceration (Definitely Related) | 0 | 0
  Malaise (Possibly Related) | 2 | 0
  Malaise (Probably Related) | 0 | 0
  Malaise (Definitely Related) | 0 | 0
  Chest discomfort (Possibly Related) | 0 | 0
  Chest discomfort (Probably Related) | 0 | 0
  Chest discomfort (Definitely Related) | 0 | 0
  Chills (Possibly Related) | 1 | 0
  Chills (Probably Related) | 0 | 0
  Chills (Definitely Related) | 0 | 0
  Dyspnoea (Possibly Related) | 0 | 0
  Dyspnoea (Probably Related) | 0 | 0
  Dyspnoea (Definitely Related) | 0 | 0
  Cough (Possibly Related) | 0 | 1
  Cough (Probably Related) | 0 | 0
  Cough (Definitely Related) | 0 | 0
  Electrocardiogram T wave abnormal (Possibly Related) | 0 | 1
  Electrocardiogram T wave abnormal (Probably Related) | 0 | 0
  Electrocardiogram T wave abnormal (Definitely Related) | 0 | 0
  Platelet count decreased (Possibly Related) | 0 | 0
  Platelet count decreased (Probably Related) | 0 | 0
  Platelet count decreased (Definitely Related) | 0 | 0
  Tachycardia (Possibly Related) | 0 | 0
  Tachycardia (Probably Related) | 0 | 0
  Tachycardia (Definitely Related) | 0 | 0
  Upper respiratory tract infection (Possibly Related) | 0 | 0
  Upper respiratory tract infection (Probably Related) | 0 | 0
  Upper respiratory tract infection (Definitely Related) | 0 | 0
  Musculoskeletal pain (Possibly Related) | 1 | 0
  Musculoskeletal pain (Probably Related) | 0 | 0
  Musculoskeletal pain (Definitely Related) | 0 | 0

21. Secondary Outcome: Number of Participants With Concomitant Medications
Description: Number of participants with concomitant medications were reported in this outcome measure.
Time Frame: From viral challenge on Day 0 up to end of follow-up (Day 28)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | RV299 | Placebo
Number analyzed (Participants) | 39 | 40
Participants | 17 | 16

22. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) for RV299
Time Frame: Pre-dose, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8,10, 12, 24, 36, 48, 60, 72, 84 and 96-hours post-dose 1 and dose 10
Population: Pharmacokinetic (PK) population consisted of all participants from ITT population (all randomized participants who received challenge virus and at least 1 dose of IMP) with at least one post-dose PK result.
Measure: Median (Full Range); unit: Hours
Arm/Group | RV299
Number analyzed (Participants) | 39
Hours
  Dose 1 | 2.85 [0.93 to 10.00]
  Dose 10 | 2.45 [0.92 to 12.13]

23. Secondary Outcome: Terminal Half-Life (t1/2) for RV299
Time Frame: Pre-dose, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8,10, 12, 24, 36, 48, 60, 72, 84 and 96 hours post-dose 1 and dose 10
Population: PK population consisted of all participants from ITT population (all randomized participants who received challenge virus and at least 1 dose of IMP) with at least one post-dose PK result. Here, 'Number Analyzed' signifies participants evaluable for specified timepoints. t1/2 for dose 1 could not be calculated as at least 3 data points were required in terminal elimination phase within same participant; this criteria could not be fulfilled due to insufficient data above limit of quantification.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | RV299
Number analyzed (Participants) | 39
Hours
  Dose 1 | NA (NA) — t1/2 for dose 1 data could not be calculated as the percentage AUC extrapolated was greater than 20% and also due to inadequate characterization of the terminal elimination phase.
  Dose 10: number analyzed (Participants) | 37
  Dose 10 | 12.1 (6.0)

24. Secondary Outcome: Maximum Observed Plasma Concentration for RV299
Time Frame: Pre-dose, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8,10, 12, 24, 36, 48, 60, 72, 84 and 96 hours post-dose 1 and dose 10
Population: PK population consisted of all participants from ITT population (all randomized participants who received challenge virus and at least 1 dose of IMP) with at least one post-dose PK result.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | RV299
Number analyzed (Participants) | 39
Nanograms per milliliter
  Dose 1 | 448 (155)
  Dose 10 | 1144 (647)

25. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to the End of the Dosing Interval for RV299
Description: Area under the plasma concentration-time curve from time zero to the end of the dosing interval for RV299 where dosing interval=12 hours.
Time Frame: Pre-dose, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8,10, 12 hours post-dose 1 and dose 10
Population: PK population consisted of all participants from ITT population (all randomized participants who received challenge virus and at least 1 dose of IMP) with at least one post-dose PK result Here, 'Number Analyzed' signifies participants evaluable for the specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | RV299
Number analyzed (Participants) | 39
Hours*nanograms per milliliter
  Dose 1: number analyzed (Participants) | 38
  Dose 1 | 3500 (825)
  Dose 10 | 7845 (3004)

26. Secondary Outcome: Area Under the Plasma Concentration-Time Curve Over the Last 24 Hours Dosing Interval for RV299
Time Frame: Pre-dose, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8,10, 12, 24 hours post-dose 1 and dose 10
Population: PK population consisted of all participants from ITT population (all randomized participants who received challenge virus and at least 1 dose of IMP) with at least one post-dose PK result. Only participants with evaluable results for this PK parameter were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | RV299
Number analyzed (Participants) | 39
Hours*nanograms per milliliter | NA (NA) — AUC24 over the dosing interval could not be computed as the dosing interval was not 24 hours.

27. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity for RV299 on Day 1
Time Frame: Pre-dose, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8,10, 12, 24, 36, 48, 60, 72, 84 and 96 hours post-dose 1
Population: PK population consisted of all participants from ITT population (all randomized participants who received challenge virus and at least 1 dose of IMP) with at least one post-dose PK result. AUC(0-infinity) could not be calculated as atleast 3 data points are required in terminal elimination phase within same participant; this criteria could not be fulfilled due to insufficient data above limit of quantification and did not include a characterization of the terminal elimination.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | RV299
Number analyzed (Participants) | 39
Hours*nanograms per milliliter | NA (NA) — Data could not be calculated as the percentage AUC extrapolated was greater than 20% and also due to inadequate characterization of the terminal elimination phase.

ADVERSE EVENTS:
Time Frame: From first dose of IMP until end of follow-up visit (up to Day 28) and from viral challenge on Day 0 up to end of follow-up (Day 28)
Arm/Group | RV299 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/40
Other Adverse Events (participants affected / at risk) | 12/39 | 12/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RV299 (N=39) | Placebo (N=40)
Headache (Nervous system disorders) | 2 | 2
Dizziness (Nervous system disorders) | 2 | 0
Ageusia (Nervous system disorders) | 0 | 1
Anosmia (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Vessel puncture site bruise (General disorders) | 1 | 2
Chills (General disorders) | 1 | 0
Malaise (General disorders) | 2 | 0
Vessel puncture site haematoma (General disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Blood potassium increased (Investigations) | 1 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Bundle branch block (Cardiac disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/91/NCT06067191/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT06067191/SAP_001.pdf